CLINICAL TRIAL: NCT02885155
Title: Contribution of Echocardiography to Prognostic Evaluation of Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2006CPRC/CHABOT
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with pulmonary arterial hypertension
  Interventions: Other: Echocardiography; Other: Hemodynamic examinations (right cardiac catheterization)

INTERVENTIONS:
Other: Echocardiography — planned at regular intervals
Other: Hemodynamic examinations (right cardiac catheterization) — planned at regular intervals

SUMMARY:
The purpose of this study is to determine the prognostic value of echocardiographic parameters in comparison with clinical and hemodynamic parameters in pulmonary arterial hypertension (PAH).

A secondary purpose of this study is to analyze the disease evolution after 3 to 6 months. In pulmonary fibrosis it has been demonstrated that the variation of clinical and paraclinical parameters between 2 examinations has a prognostic interest. In this study the prognostic value of variation of some echocardiographic parameters between initial examination and echocardiography after 3 or 6 months will be evaluated.

Another secondary purpose is to create a common database for Pneumology, Cardiology and Epidemiology departments with prospective registration of new cases of PAH and follow of patients under treatment.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a rare pathology with a poor prognosis and a median survival lower than 3 years in the absence of a specific treatment.

The prognostic evaluation is based on clinical and hemodynamic data needing the right cardiac catheterization. It has been shown that prognosis depends essentially on the severity of right ventricular dysfunction. Recently, various echocardiographic parameters derived from new techniques such as tissue Doppler have been validated for the evaluation of right ventricular function. Some have been used as prognostic factor in cardiac insufficiency, but not in PAH.

This is an observational retrospective and then prospective study. Usual PAH assessment includes a complete clinical and paraclinical evaluation. History and physical examination assess dyspnea, search signs of disease severity and quantify functional impact of 6 min-walking test. An echocardiography and a right cardiac catheterization are realized in all patients. Clinical consultations of patients and control echocardiographic and hemodynamic examinations are programmed at regular intervals.

The demonstration of prognostic value of some echocardiographic parameters could diminish right cardiac catheterizations.

ELIGIBILITY:
Inclusion Criteria:

* Mean pulmonary artery pressure > 25 mmHg in hemodynamics
* according to Venice classification: Idiopathic PAH or associated to other known risk factors (anorectics, portal hypertension, connective tissue diseases, in particular scleroderma but also lupus, congenital heart disease with Eisenmenger syndrome, HIV infection)

Exclusion Criteria:

* Atrial fibrillation
* Poor echogenicity
* PAH associated to another factor, thromboembolic disease, respiratory insufficiency, left heart disease or mitral or aortic valvulopathy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary arterial hypertension followed at CHU Nancy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Mortality at 5 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: François Chabot, Pr, Principal Investigator — Service de Maladies Respiratoires et Réanimation Respiratoire - CHU Nancy

IPD SHARING:
Plan to Share IPD: No